CLINICAL TRIAL: NCT05630508
Title: mHealth Lifestyle Management Program (LIVEN) For Adults With Diabetes Type 2: A Feasibility Study
Brief Title: Lifestyle Management App for Adults With Diabetes Type
Acronym: LIVEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Liven (Unknown)
Responsible Party: Principal Investigator, Shaima Alothman, Research Scientist, Clinical Assistant Professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-0140
Record Dates: First submitted 2022-10-10; First posted 2022-11-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes management; Mhealth lifestyle management program
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: The participant won't know if they got the full or sham or no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- interactive mhealth Lifestyle behavior intervention (Experimental): Receiving Standard care, LIVEN educational material and interactive LIVEN application
  Interventions: Behavioral: interactive Mhealth Lifestyle behavior intervention
- Sham group - app access only (Sham Comparator): Receiving standard care, LIVEN educational material and access to the application
  Interventions: Other: Sham
- Control group - Standard care (No Intervention): Receiving Standard care only

INTERVENTIONS:
Behavioral: interactive Mhealth Lifestyle behavior intervention — Receiving Standard care, LIVEN educational material and interactive LIVEN application, via having a human component which is a health coach for 3 months
  Arms: interactive mhealth Lifestyle behavior intervention
Other: Sham — Receiving standard care, LIVEN educational material and access to the application
  Arms: Sham group - app access only

SUMMARY:
This study will evaluate whether the 12-week health coaching mobile application (LIVEN) will succeed in enhancing lifestyle behaviors in adults with Type 2 Diabetes compared to typical treatment. The mobile application's viability will be assessed in 2 parts; the first part is testing easiness and friendliness of using Liven by the patient and health coach. The second part is evaluating the suitability of Liven education material for the patients and whether the coaching program results in enhancing lifestyle behaviors and blood sugar levels. the investigators hypothesize that the 12-week online lifestyle-coaching program will be viable, and a full-scale study can proceed.

DETAILED DESCRIPTION:
This study will investigate the feasibility of a 12-weeks online lifestyle (nutrition and physical behavior) coaching program through a mobile app (LIVEN) compared to standard treatment for people with type 2 diabetes. This study will be done in two phases; the first phase is the usability study (phase1), in which the user friendliness of the application will be assessed, and any technical flaws will be resolved prior and during the second phase. The second phase of the study will consist of adapting a diabetes educational material and assessing the feasibility of the program (phase2). the investigators hypothesize that the 12-week online lifestyle-coaching program will be feasible, and a full-scale study can proceed.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18 years or older
* Arabic speakers
* Capable of utilizing smartphones
* Diagnosed with T2DM
* Poor glycemic control: A1c > 7.5%

Exclusion Criteria:

* Individuals using insulin injection
* Individuals suffering from disorders that might affect intervention (e.g. amputation, enucleation of the eye, or end-stage kidney disease)
* Women who are pregnant or breastfeeding
* Individuals diagnosed with other types of diabetes (such as type I or MODY)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
recruitment rate - descriptive | immediately after the intervention (3 months)
  reported as the number of participants' consented divide by the number of people that were invited to participate
retention rates | immediately after the intervention (3 months)
  reported as the number of participants completing all study sessions
User friendliness | Daily application engagement data for each patient will be analyzed once at the end of the patient's 12 week program.
  will be assessed via user engagement tracking in the app

SECONDARY OUTCOMES:
Glycemic control - A1c | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assess via A1c blood test will be reported as percentage. higher % indicate worse outcome
Glycemic control - continuous glucose mentoring (CGM) | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assess via continuous glucose mentoring (CGM) as variability. higher variability indicates worse outcome
Body composition - fat free mass (%) physiological parameter | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assessed via Bioelectrical Impedance Analysis (BIA). fat free mass (%) will reported as percentage. higher % indicate better outcome
Lifestyle behaviors - Health-Promoting Lifestyle profile II (Questionnaire) | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assessed via Health-Promoting Lifestyle profile II. HPLP-II is a 4-point Likert scale with 52 items including six subscales: health responsibility, physical activity, nutrition, spiritual growth, interpersonal relationships, and stress management. scores range from 52 to 208. higher scores indicate better outcome.
physical performance assessments - upper body muscle strength in kg | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assessed via Hand Grip Strength using dynameter (power in kg), higher scores indicate higher physical performance
physical performance assessments - lower body muscle strength in counts | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assessed via Sit to Stand Test (count), higher counts indicate higher physical performance
physical performance assessments - endurance | will be assessed one week prior to the intervention and one week after the end of the intervention
  will be assessed via 6-minute walk test (distance in m). higher distance indicates higher endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Nourah bint Abdulrahman University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided